CLINICAL TRIAL: NCT05952518
Title: Evaluation of Peripheral Nerve Stimulation as an Alternative to Radiofrequency Ablation for Facet Joint Pain
Brief Title: PNS vs RFA for Facet Joint Pain
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants have been enrolled to date. The study is currently under consideration for early termination due to recruitment challenges.
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Daniel Cortes, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022997
Record Dates: First submitted 2023-06-15; First posted 2023-07-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Facet Joint Pain
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Peripheral Nerve Stimulation (Experimental): Peripheral nerve stimulation (PNS) is a procedure used to relieve chronic back pain by targeting the nerves responsible for transmitting pain signals from the back to the brain. It is a minimally invasive approach that aims to disrupt the pain signals and provide pain relief.
  Interventions: Device: Sprint PNS system
- Radiofrequency Ablation (Active Comparator): Radiofrequency ablation (RFA) is the current standard of care for facet joint pain. It is a minimally invasive procedure used to relieve chronic back or neck pain caused by issues with the small joints in the spine called facet joints.
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Device: Sprint PNS system — Temporary electrical stimulation of the medial nerve with implanted wires and wearable stimulator
  Arms: Peripheral Nerve Stimulation
Procedure: Radiofrequency Ablation — Thermal ablation of the medial nerve
  Arms: Radiofrequency Ablation

SUMMARY:
Radiofrequency ablation of the medial nerve is the current surgical treatment for back pain originating from the facet joints in the spine. However, this procedure causes denervation of spinal muscles. Peripheral nerve stimulation is another treatment for facet joint pain that may not cause damage to the spinal muscles. This study will compare both treatments in terms pain relief and spine biomechanics.

ELIGIBILITY:
Inclusion Criteria:

1. Age range (18-80 years): The age range of the patient population at Hershey Medical Center with facet pain is 24 to 90 years old, with a mean age of 63 years old. Due to the physical tests planned in the study, the maximum age limit will be restricted to 80 years old.
2. English Speaking: Adults who only speak other languages will not be included because of the lack of feasibility of employing reliable instruments and interviewers fluent in other languages.
3. Facet Joint Pain: male and female patients having a diagnosis of facet joint pain based upon accepted diagnostic criteria (i.e., two positive nerve blocks) and assessed by an experienced physical therapist or physician.
4. Indication for Surgical Procedure: Physical therapy is the first line of action for facet joint pain. If PT is not effective, patients are eligible for RFA or PNS.

Exclusion Criteria:

1. Previous Spinal Conditions Surgery: We will exclude patients with other spinal conditions like scoliosis or who have received previous spinal surgeries.
2. Systemic neurological or neuromuscular disease: Such disorders (e.g., stroke, muscular dystrophy, myopathies) affect muscle and may confound muscle data and/or balance and physical performance data.
3. Allergic reaction to ultrasound gels: It is possible, although rare, that patients develop allergic reaction to ultrasound gels. Those subjects will be excluded from the study.
4. Physical Activity: Subjects will be asked to fill out the Physical Activity Readiness Questionnaire (PAR-Q), and if they answer yes to any of the questions, they need to be cleared by their physician prior to participating in the study.
5. Current infection, illness, or condition: Individuals with a current infection, illness, or condition (e.g., uncontrolled blood pressure, pregnancy) that may affect their ability to safely participate will be excluded.
6. Mental incompetency: Individuals who cannot legally consent themselves to the surgical procedure and participation in the research study, will not be considered for inclusion.
7. Patients who have a Deep Brain Stimulation (DBS) system.
8. Patients who have an implanted active cardiac implant (e.g. pacemaker or defibrillator).
9. Patients who have any other implantable neuro-stimulator whose stimulus current pathway may overlap with that of the SPRINT System.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Multifidus muscle activity | pre-treatment
  Muscle contraction quantification via shear wave elastography
Multifidus muscle activity | within two weeks of treatment completion
  Muscle contraction quantification via shear wave elastography
Multifidus muscle activity | 12 months after pre-treatment measurement
  Muscle contraction quantification via shear wave elastography

SECONDARY OUTCOMES:
Pain Intensity | pre-treatment
  Visual Analog Scale, scale range 1 - 10, 10 being worse possible pain.
Pain Intensity | within two weeks of treatment completion
  Visual Analog Scale, scale range 1 - 10, 10 being worse possible pain.
Pain Intensity | 12 months after pre-treatment measurement
  Visual Analog Scale, scale range 1 - 10, 10 being worse possible pain.
Oswestry Disability Index | pre-treatment
  Survey evaluating disability level, 0 - 4 No disability 5 - 14 Mild disability 15 - 24 Moderate disability 25 - 34 Severe disability 35 - 50 Completely disabled
Oswestry Disability Index | within two weeks of treatment completion
  Survey evaluating disability level, 0 - 4 No disability 5 - 14 Mild disability 15 - 24 Moderate disability 25 - 34 Severe disability 35 - 50 Completely disabled
Oswestry Disability Index | 12 months after pre-treatment measurement
  Survey evaluating disability level, 0 - 4 No disability 5 - 14 Mild disability 15 - 24 Moderate disability 25 - 34 Severe disability 35 - 50 Completely disabled
PROMIS-29 v2.0 | pre-treatment
  Survey assessing pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance)
PROMIS-29 v2.0 | within two weeks of treatment completion
  Survey assessing pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance)
PROMIS-29 v2.0 | 12 months after pre-treatment measurement
  Survey assessing pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance)
isometric back strength | pre-treatment
  Measurement of peak force generated by the torso in extension in Newtons
Isometric back strength | within two weeks of treatment completion
  Measurement of peak force generated by the torso in extension in Newtons
isometric back strength | 12 months after pre-treatment measurement
  Measurement of peak force generated by the torso in extension in Newtons
Functional Reach | pre-treatment
  distance between the length of an outstretched arm in a maximal forward reach, 10"/25 cm or greater Low risk of falls, 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal, 6"/15cm or less Risk of falling is 4x greater than normal, Unwilling to reach Risk of falling is 8x greater than normal.
Functional Reach | within two weeks of treatment completion
  distance between the length of an outstretched arm in a maximal forward reach, 10"/25 cm or greater Low risk of falls, 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal, 6"/15cm or less Risk of falling is 4x greater than normal, Unwilling to reach Risk of falling is 8x greater than normal.
Functional Reach | 12 months after pre-treatment measurement
  distance between the length of an outstretched arm in a maximal forward reach, 10"/25 cm or greater Low risk of falls, 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal, 6"/15cm or less Risk of falling is 4x greater than normal, Unwilling to reach Risk of falling is 8x greater than normal.
Repetitive Trunk Rotation | pre-treatment
  Time to complete 20 rotations, seconds, longer times are worse performance.
Repetitive Trunk Rotation | within two weeks of treatment completion
  Time to complete 20 rotations, seconds, longer times are worse performance.
Repetitive Trunk Rotation | 12 months after pre-treatment measurement
  Time to complete 20 rotations, seconds, longer times are worse performance.
Repeated Chair Stands | pre-treatment
  Time to perform 5 repeated chair stands, higher times mean worse outcomes.
Repeated Chair Stands | within two weeks of treatment completion
  Time to perform 5 repeated chair stands, higher times mean worse outcomes.
Repeated Chair Stands | 12 months after pre-treatment measurement
  Time to perform 5 repeated chair stands, higher times mean worse outcomes.
Pfirmmann grade | pre-treatment
  Degeneration of lumbar discs at the treated level, grade 1 - 5, 1 is normal and 5 is completely collapsed disc.
Pfirmmann grade | within two weeks of treatment completion
  Degeneration of lumbar discs at the treated level, grade 1 - 5, 1 is normal and 5 is completely collapsed disc.
Pfirmmann grade | 12 months after pre-treatment measurement
  Degeneration of lumbar discs at the treated level, grade 1 - 5, 1 is normal and 5 is completely collapsed disc.
t2-relaxation time | pre-treatment
  T2 relaxation time of the disc at the treated level. Lower values indicate more degeneration.
t2-relaxation time | within two weeks of treatment completion
  T2 relaxation time of the disc at the treated level. Lower values indicate more degeneration.
t2-relaxation time | 12 months after pre-treatment measurement
  T2 relaxation time of the disc at the treated level. Lower values indicate more degeneration.
2-point dixon MRI | pre-treatment
  Intramuscular fat percentage, higher percentage means worse outcome.
2-point dixon MRI | within two weeks of treatment completion
  Intramuscular fat percentage, higher percentage means worse outcome.
2-point dixon MRI | 12 months after pre-treatment measurement
  Intramuscular fat percentage, higher percentage means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Cortes, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided